CLINICAL TRIAL: NCT01178736
Title: Efficacy of a Combined Program for Early Detection of Breast and Gynecological Cancers in Low Resource Countries
Brief Title: Early Detection of Cancers in Low Resource Countries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Woman's Cancer Foundation (Other)
Responsible Party: Mahesh Shetty, MD/President, Woman's Cancer Foundation
Other Study IDs: WCF-2011-BRA-IND-CAM
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms
Keywords: neoplasms
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Screening and Diagnosis: Screening of asymptomatic women for Breast and Cervical cancer in the age group of 35-64 years. Diagnostic assessment of symptomatic women for Ovarian and Endometrial cancer in the age group of 50-64 years.
  Interventions: Procedure: Breast Cancer Screening and Diagnosis; Procedure: Cervical Cancer Screening and Diagnosis; Procedure: Ovarian Cancer Screening and Diagnosis; Procedure: Endometrial Cancer Screening and Diagnosis

INTERVENTIONS:
Procedure: Breast Cancer Screening and Diagnosis — Clinical Breast Examination and Sonography followed by Fine needle aspiration biopsy (FNAB) of screen positive cases.
  Other Names: FNAB; CBE; Ultrasound
Procedure: Cervical Cancer Screening and Diagnosis — Visual Inspection with Acetic acid, PAP smear or Human Papilloma Virus DNA testing followed by Cryotherapy of screen positive cases.
  Other Names: HPV DNA
Procedure: Ovarian Cancer Screening and Diagnosis — Transvaginal sonogram and clinical evaluation in post menopausal women with symptoms suggestive of ovarian cancer.
  Other Names: Ultrasound
Procedure: Endometrial Cancer Screening and Diagnosis — Transvaginal sonographic assessment of the endometrial stripe in post menopausal women with abnormal bleeding.
  Other Names: Ultrasound

SUMMARY:
The purpose of this study is to implement a community-based combined program for early detection of breast, cervical, ovarian and endometrial cancer in low-resource countries delivered through a free standing or a mobile Well Woman Clinic. The goals of this program are to downstage cancers and improve mortality rates using low-cost early detection methods. These programs will be implemented in regions where early cancer detection strategies are not in place and cancers present at advanced stages with resultant high mortality. Currently, there are three target project sites: Cambodia (June 2011), India (June 2011), and Brazil (March 2011). Memorandums of Understanding have been secured with local health organizations in each region to establish clinic operations. Each clinic would serve an approximate target population of 100,000 amongst whom about 12,000 eligible women (4-5,000 annually) will be invited to be screened for breast and cervical cancer over a three-year time span.

DETAILED DESCRIPTION:
We will study the use of sonographic screening in addition to Clinical Breast Examination in low resource settings where screening programs are not currently in place and establishing a population based mammographic screening would be expensive, resource intensive, and difficult if not impossible to implement. The effectiveness of the screening and diagnostic methodology used for early detection of breast, cervical, ovarian and endometrial cancers in low resource settings will be studied. The program would involve screening of asymptomatic women for Breast and Cervical cancer and diagnostic assessment of symptomatic women for Ovarian and Endometrial cancer. Women in the age group of 30-59 yrs will be screened once every three years utilizing the following methods: Breast - clinical breast examination [CBE] and Sonography, followed by Fine needle aspiration biopsy (FNAB) of screen positive cases; Cervical - Human Papilloma Virus DNA testing followed by Cryotherapy of screen positive cases (Single visit, screen and treat approach); Ovarian - Transvaginal sonogram and clinical evaluation; Endometrial - Transvaginal sonographic assessment of the endometrial stripe.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer: women age 35-64
* Cervical Cancer: women age 30-59
* Ovarian Cancer: symptomatic post menopausal women age 50-64
* Endometrial Cancer: symptomatic post menopausal women age 50-64

Exclusion Criteria:

* women under the age of 30

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Brazil has two rural hospitals serving a population of roughly 46,000 people (Nova Andradina) inside Mato Grosso do Sul, which has a population of over 2 million. Cambodia has a population of over 1 million inside the Phnom Penh metropolitan area. India has a population of more than 1.3 million inside the state of Goa. According to the NFHS-2, nearly 30 percent of rural Goan women live 10 or more kilometers away from a primary health center.
Sampling Method: Non-Probability Sample
Enrollment: 36000 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The Effectiveness of an Innovative, Low-Cost Screening and Diagnostic Methodology | Three (3) year interval
  This study will examine the effectiveness of an innovative, low-cost screening and diagnostic methodology used for combined early detection of breast and gynecological cancers in low resource regions where early cancer detection strategies are not in place and cancers currently are diagnosed at advanced stages with resultant high mortality.

SECONDARY OUTCOMES:
Effectiveness of CBE and Ultrasonography for Breast Cancer Detection | Three (3) year interval
  This study will examine the effectiveness of Clinical Breast Examination combined with Ultrasonography for breast cancer screening and detection in low resource settings where X-ray mammography proves not feasible in terms of cost, technology, and staff.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Yang, MD, Principal Investigator — M.D. Anderson Cancer Center, University of Texas; Diljeet K Singh, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Adhemar Longatto Filho, MD, Principal Investigator — University of Sao Paolo
Locations (3):
- Hospital de Cancer de Barretos, São Paulo, Brazil
- Sihanouk Hospital Center of Hope, Hope Worldwide Cambodia, Phnom Penh, Cambodia
- Manipal Healthcare Group, Goa, India

REFERENCES:
- [Background] Elmore JG, Armstrong K, Lehman CD, Fletcher SW. Screening for breast cancer. JAMA. 2005 Mar 9;293(10):1245-56. doi: 10.1001/jama.293.10.1245. PMID 15755947
- [Background] Kuhl CK. The "coming of age" of nonmammographic screening for breast cancer. JAMA. 2008 May 14;299(18):2203-5. doi: 10.1001/jama.299.18.2203. No abstract available. PMID 18477789
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Background] Kolb TM, Lichy J, Newhouse JH. Comparison of the performance of screening mammography, physical examination, and breast US and evaluation of factors that influence them: an analysis of 27,825 patient evaluations. Radiology. 2002 Oct;225(1):165-75. doi: 10.1148/radiol.2251011667. PMID 12355001
- [Background] Kaplan SS. Clinical utility of bilateral whole-breast US in the evaluation of women with dense breast tissue. Radiology. 2001 Dec;221(3):641-9. doi: 10.1148/radiol.2213010364. PMID 11719658
- [Background] Tohno E, Ueno E, Watanabe H. Ultrasound screening of breast cancer. Breast Cancer. 2009;16(1):18-22. doi: 10.1007/s12282-008-0082-8. Epub 2008 Nov 14. PMID 19009372
- [Background] Sankaranarayanan R, Nene BM, Shastri SS, Jayant K, Muwonge R, Budukh AM, Hingmire S, Malvi SG, Thorat R, Kothari A, Chinoy R, Kelkar R, Kane S, Desai S, Keskar VR, Rajeshwarkar R, Panse N, Dinshaw KA. HPV screening for cervical cancer in rural India. N Engl J Med. 2009 Apr 2;360(14):1385-94. doi: 10.1056/NEJMoa0808516. PMID 19339719
- [Background] Schiffman M, Wacholder S. From India to the world--a better way to prevent cervical cancer. N Engl J Med. 2009 Apr 2;360(14):1453-5. doi: 10.1056/NEJMe0901167. No abstract available. PMID 19339726
- [Background] Goldie SJ, Kuhn L, Denny L, Pollack A, Wright TC. Policy analysis of cervical cancer screening strategies in low-resource settings: clinical benefits and cost-effectiveness. JAMA. 2001 Jun 27;285(24):3107-15. doi: 10.1001/jama.285.24.3107. PMID 11427139
- [Background] Goff BA, Mandel LS, Drescher CW, Urban N, Gough S, Schurman KM, Patras J, Mahony BS, Andersen MR. Development of an ovarian cancer symptom index: possibilities for earlier detection. Cancer. 2007 Jan 15;109(2):221-7. doi: 10.1002/cncr.22371. PMID 17154394
- [Background] Goff BA, Mandel LS, Melancon CH, Muntz HG. Frequency of symptoms of ovarian cancer in women presenting to primary care clinics. JAMA. 2004 Jun 9;291(22):2705-12. doi: 10.1001/jama.291.22.2705. PMID 15187051
- [Background] Menon U, Gentry-Maharaj A, Hallett R, Ryan A, Burnell M, Sharma A, Lewis S, Davies S, Philpott S, Lopes A, Godfrey K, Oram D, Herod J, Williamson K, Seif MW, Scott I, Mould T, Woolas R, Murdoch J, Dobbs S, Amso NN, Leeson S, Cruickshank D, McGuire A, Campbell S, Fallowfield L, Singh N, Dawnay A, Skates SJ, Parmar M, Jacobs I. Sensitivity and specificity of multimodal and ultrasound screening for ovarian cancer, and stage distribution of detected cancers: results of the prevalence screen of the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS). Lancet Oncol. 2009 Apr;10(4):327-40. doi: 10.1016/S1470-2045(09)70026-9. Epub 2009 Mar 11. PMID 19282241
- [Background] van Nagell JR Jr, DePriest PD, Ueland FR, DeSimone CP, Cooper AL, McDonald JM, Pavlik EJ, Kryscio RJ. Ovarian cancer screening with annual transvaginal sonography: findings of 25,000 women screened. Cancer. 2007 May 1;109(9):1887-96. doi: 10.1002/cncr.22594. PMID 17373668
- [Background] Van den Bosch T, Van Schoubroeck D, Domali E, Vergote I, Moerman P, Amant F, Timmerman D. A thin and regular endometrium on ultrasound is very unlikely in patients with endometrial malignancy. Ultrasound Obstet Gynecol. 2007 Jun;29(6):674-9. doi: 10.1002/uog.4031. PMID 17523157
- [Background] Smith-Bindman R, Kerlikowske K, Feldstein VA, Subak L, Scheidler J, Segal M, Brand R, Grady D. Endovaginal ultrasound to exclude endometrial cancer and other endometrial abnormalities. JAMA. 1998 Nov 4;280(17):1510-7. doi: 10.1001/jama.280.17.1510. PMID 9809732
- [Background] Tabor A, Watt HC, Wald NJ. Endometrial thickness as a test for endometrial cancer in women with postmenopausal vaginal bleeding. Obstet Gynecol. 2002 Apr;99(4):663-70. doi: 10.1016/s0029-7844(01)01771-9. PMID 12039131
- [Background] Amant F, Moerman P, Neven P, Timmerman D, Van Limbergen E, Vergote I. Endometrial cancer. Lancet. 2005 Aug 6-12;366(9484):491-505. doi: 10.1016/S0140-6736(05)67063-8. PMID 16084259